CLINICAL TRIAL: NCT04782284
Title: Effect of Comprehensive Swallowing Rehabilitation in Patients With Multiple System Atrophy: A Randomized Controlled Trial
Brief Title: Comprehensive Swallowing Rehabilitation in Patients With MSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Han Gil Seo, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MSA-swrehab-RCT
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Multiple System Atrophy
Keywords: Multiple System Atrophy; Dysphagia; Swallowing rehabilitation; Videofluoroscopic Swallowing Study
MeSH Terms: conditions — Multiple System Atrophy; Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Comprehensive swallowing rehabilitation (Experimental)
  Interventions: Other: Comprehensive swallowing rehabilitation
- Swallowing education (Active Comparator)
  Interventions: Other: Swallowing education

INTERVENTIONS:
Other: Comprehensive swallowing rehabilitation — The treatment time per session is 30 minutes. Total 12 sessions are provided for 6 weeks.
  Arms: Comprehensive swallowing rehabilitation
Other: Swallowing education — The education is 30 minutes. Total 1 session is provided immediately after baseline evaluation.
  Arms: Swallowing education

SUMMARY:
The purpose of this study is to investigate the effect of comprehensive swallowing rehabilitation in patients with multiple system atrophy.

DETAILED DESCRIPTION:
Multiple system atrophy (MSA) is a rapidly progressive neurodegenerative disease characterized by parkinsonism, cerebellar syndrome, and autonomic failure. Dysphagia is a clinically significant symptom leading to pneumonia that causes death in patients with MSA. Although the symptoms of dysphagia in the two subtypes of MSA-the parkinsonian variant and the cerebellar variant- are different, there is no significant difference in the latency to onset of tube feeding. Therefore, effective intervention is needed to improve the safety and efficiency of swallowing regardless of the subtypes of MSA.

Although swallowing rehabilitation has been widely applied for swallowing disorders in patients with MSA, few studies have reported the clinical effect of applying swallowing therapy. Comprehensive swallowing rehabilitation has focused on functional muscle training, compensatory swallowing maneuvers, and thermal-tactile stimulation, which is used to treat dysphagia from stroke, Parkinson's disease, and head and neck cancer. Therefore, this study aims to investigate the effect of comprehensive swallowing rehabilitation in patients with MSA.

ELIGIBILITY:
Inclusion Criteria:

* Age >19 years
* Clinically diagnosed with MSA according to the guidelines of the 2nd consensus of the Gilman criteria
* Clinically diagnosed to have dysphagia by a physiatrist
* Two or more points on the Penetration-aspiration scale (PAS) from the Videofluoroscopic swallowing study (VFSS) conducted within 3 months

Exclusion Criteria:

* Moderate to severe cognitive dysfunction with Mini-mental State Examination score < 19
* Comorbidities or structural abnormalities that may affect swallowing function
* Other comorbidities that make it difficult to participate in the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-05-17 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Penetration-Aspiration Scale | at 6 weeks
Videofluoroscopic dysphagia scale | at 6 weeks

SECONDARY OUTCOMES:
Penetration-Aspiration Scale | at 12 weeks
Videofluoroscopic dysphagia scale | at 12 weeks
Peak Cough Flow | at 6 weeks, at 12 weeks
Maximal Inspiratory Pressure | at 6 weeks, at 12 weeks
Maximal Expiratory Pressure | at 6 weeks, at 12 weeks
Forced vital capacity | at 6 weeks, at 12 weeks
Forced expiratory volume | at 6 weeks, at 12 weeks
Maximal phonation time | at 6 weeks, at 12 weeks
Swallowing disturbance questionnaire | at 6 weeks, at 12 weeks
Swallowing Quality of Life questionnaire | at 6 weeks, at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Han Gil Seo, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No